CLINICAL TRIAL: NCT05568108
Title: Using the Masseteric Nerve for Facial Nerve Reanimation: A Clinical Study.
Brief Title: Using the Masseteric Nerve for Facial Nerve Reanimation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Refaat Ahmed Abdelkarim, assitant lecturer of plastic and reconstructive surgery, Assiut University
Other Study IDs: Masseteric for facial nerve
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Facial Nerve Paresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- nerve transfer: masseteric nerve to central branch facial nerve. (Early fibrillation on EMG)
  Interventions: Procedure: masseteric nerve to central branch facial nerve
- nerve and free functioning muscle transfer: Masseteric nerve to free functioning muscle transfer. (Late no fibrillation on EMG)
  Interventions: Procedure: Masseteric nerve to free functioning muscle transfer

INTERVENTIONS:
Procedure: masseteric nerve to central branch facial nerve — masseteric nerve to central branch facial nerve. (Early fibrillation on EMG)
  Groups: nerve transfer
Procedure: Masseteric nerve to free functioning muscle transfer — Masseteric nerve to free functioning muscle transfer. (Late no fibrillation on EMG)
  Groups: nerve and free functioning muscle transfer

SUMMARY:
The return of eyelid function and facial expression in Patients with facial nerve affection is very important for quality of life. Eyelid dysfunction leads to drying and ulceration of cornea which may lead to permanent vision loss.

Facial paralysis is distinguished into two main groups according to the presence or absence of facial fibrillations at needle Electromyography. Recent paralysis, mainly lasting less than two years generally show these signs and are eligible for reactivation of facial nerve by anastomosing it to a donor one (early facial reanimation).

The masseteric nerve (motor branch of trigeminal nerve ) is a reliable donor nerve on early facial reanimation So on this study we examine the advantages and disadvantages of using masseteric nerve to develop a protocol for use of facial reanimation and restoration of function on facial paresis.

DETAILED DESCRIPTION:
Type of the study: observtional Study (clinical trial)

Intervention Model Description:

Patients will be two groups according to the surgical procedure performed as follows:

* Group A: masseteric nerve to central branch facial nerve. (Early fibrillation on EMG)
* Group B: Masseteric nerve to free functioning muscle transfer. (Late no fibrillation on EMG)

Allocation and Randomization:

Twenty-four patients will be assigned to Group A early or Group B late (2 groups). group A will be for early and be will be for late cases

Study Setting: Plastic and Reconstructive Surgery Department, Assuit University Hospital and San Paolo university hospital of Milano university.

Study subjects:

Inclusion criteria:

1.Facial nerve affection 2.Patients are generally fit with no other disease interfere with microsurgery. 3.Electromyography showing fibrillations for group A and no fibrillation for group B.

b. Exclusion criteria:

1.Patient with other medical or mental disease-causing generalized paralysis. 2.Syndromic cases. 3.Patients are generally unfit or with any disease interfere with microsurgery.

c. Sample Size Calculation: 24 Sample size was calculated using G power program version 3.1.9.4 (6) in order to detect a significant difference in mean of EFACE score (one of main assessed outcomes in the study ) between two groups under the study , assumed effect size 0.6 based on clinical assumption ( novel study ), α error 0.3 , power 0.80, and allocation ratio 1: 1.

Twenty-two patient plus 10% for dropouts to make total twenty-four (12 patient for every group).

Study tools

All patients in this study are subjected to:

Pre-operative Assessment:

1. Patient history.
2. All patients will do preoperative clinical and neurophysiological assessments of mimetic muscle function and donor nerve status (the ipsilateral deep temporal nerve. The neurophysiological tests will include needle Electromyography (EMG) for recruitment of residual motor unit action potential to determine which procedure
3. The trigeminal motor component will be tested by palpating the temporalis muscle and masseteric muscle during chewing and via needle EMG to verify availability as a donor motor nerve.
4. Photographic documentation preoperative using standardized EFACE view.
5. Ophthalmological assessment of the affected eye for detection of redness, ulcer, etc.

Surgical procedure:

Group A the investigators will avoid the use of muscle relaxants to induce anaesthesia and employ an electro-stimulator to identify the masseteric nerve and the facial nerve branches supplying the affected side.

Exploration on the affected side a facelift-type incision will be performed, and an anterior subcutaneous flap is then will be lifted for several centimetres. In the inferior zygomatic region, the plane of elevation is deepened into the sub-SMAS plane and a composite flap elevated for several centimetres. Following elevation in this plane, the distal facial nerve branches will be identified. The distal portion of the zygomatic nerve is usually located midway between the oral commissure and the helical root. and was confirmed by nerve stimulator.

Then masseteric nerve identified in masseteric muscle and then end to end anastomosis with the central branch of facial nerve Then suction drain will be put and will be removed after 24 hours. Group B The same technique of face lift and harvest the free functioning muscle flap and micro anastomosis of the flap for the superficial temporal system or the facial artery system and the same technique for masseteric nerve identification and end to end anastomosis and to side for prepare cross nerve form the stage one Post-operative All patient will receive physiotherapy and post-operative follow up to detect any wound complication.

Evaluation (After 6 months from the operation)

1. Photo documentation for EFACE
2. Donor site morbidity.
3. Onset of first movement
4. Patient satisfaction

Complications:

1. General surgical complication.
2. General complication due to general anaesthesia.
3. Specific complication:

   1. Delayed healing of nerve anastomosis.
   2. Affection of mastication.
   3. No postoperative improvement.

Research outcome measures:

a. Primary (main): Comparing the outcomes on EFACE score

Secondary (subsidiary):

1. Easy technique for rapid masseteric nerve identification.
2. Effect of addition of contracted growth factor around the anastomosis
3. Procedure-related morbidity and mortality.
4. Effect of selective neurectomy for overactive affected branches with the total reanimation
5. The experience of adding another neural impots with masseteric nerve
6. Operative time and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

1. Facial nerve affection
2. Patients are generally fit with no other disease interfere with microsurgery.
3. Electromyography showing fibrillations for group A and no fibrillation for group B.

Exclusion Criteria:

1. Patient with other medical or mental disease-causing generalized paralysis.
2. Syndromic cases.
3. Patients are generally unfit or with any disease interfere with microsurgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Facial nerve affection patients
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2020-11-04 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Comparing the outcomes on EFACE score | up to one year
  difference on the score

SECONDARY OUTCOMES:
Effect of addition of contracted growth factor around the anastomosis | up to one year
  time for nerve activation

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M refaat, mcch, Principal Investigator — faculty of medcine assiut University
Locations (1):
- Plastic Surgery Department Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided